CLINICAL TRIAL: NCT03177811
Title: Effect of Acetazolamide on Postural Control in Patients With Chronic Obstructive Pulmonary Disease at Altitude: A Randomized, Placebo-controlled, Double-blind Parallel Trial
Brief Title: Effect of Acetazolamide on Postural Control in Patients With Respiratory Disease at Altitude
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2017-00137B
Record Dates: First submitted 2017-05-23; First posted 2017-06-06 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: postural control; balance performance; airway disease; altitude; prevention; acetazolamide
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACETAZOLAMIDE oral capsule (Active Comparator): Acetazolamide 375mg/day (capsule @125 mg: 1 in the morning, 2 in the evening), orally. Medication starts 24 hours before ascent to 3200m until the morning after the second night at 3200m
  Interventions: Drug: ACETAZOLAMIDE oral capsule
- PLACEBO oral capsule (Placebo Comparator): Placebo (capsules identically looking as acetazolamide capsules: 1 in the morning, 2 in the evening), orally. Medication starts 24 hours before ascent to 3200m until the morning after the second night at 3200m.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: ACETAZOLAMIDE oral capsule — Administration of 125mg acetazolamide in the morning, 250mg in the evening, starting 24 hours before departure to 3200m
  Arms: ACETAZOLAMIDE oral capsule
Drug: Placebo oral capsule — Administration of equally looking placebo capsules in the morning and evening, starting 24 hours before departure to 3200m
  Arms: PLACEBO oral capsule

SUMMARY:
In this trial, the investigators will evaluate the effect of acetazolamide (375 mg per day) vs. placebo on postural control at acute altitude exposure in patients with COPD.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind parallel trial evaluating the effect of acetazolamide (375 mg per day) vs. placebo on postural control at altitude (Tuja Ashu, 3200 m). Participants living in the Bishkek area, Kyrgyzstan (760m), will be transferred by car within 4h to the Tuja Ashu high altitude clinic (3200 m), and stay there for 2 days. Acetazolamide 375mg/day (or placebo) will be administered 24 hours before departure at 760 m and during the stay at altitude. Outcomes will be assessed during the stay at 3200 m. Randomization to acetazolamide or placebo will be carried out after baseline measurements in Bishkek (760 m).

Postural control will be assessed by a rectangular, stable balance platform (Wii Balance Board) measuring the body's center of gravity. The movement of the body's center of gravity will be recorded in a two-dimensional coordinate system and indicated as path length.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, age 18-75 yrs.
* COPD diagnosed according to GOLD, FEV1 40-80% predicted, SpO2 ≥92% at 750 m.
* Born, raised and currently living at low altitude (<800m).
* Written informed consent.

Exclusion Criteria:

* COPD exacerbation, very severe COPD with hypoxemia at low altitude (FEV1/FVC <0.7, FEV1 <40% predicted, oxygen saturation on room air <92% at 750 m).
* Comorbidities such as uncontrolled cardiovascular disease, i.e., unstable systemic arterial hypertension, coronary artery disease; previous stroke; OSA; pneumothorax in the last 2 months.
* Internal, neurologic, rheumatologic or psychiatric disease including current heavy smoking (>20 cigarettes per day)
* Known renal failure or allergy to acetazolamide and other sulfonamides

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-08-02 (Actual)

PRIMARY OUTCOMES:
Change in postural control | Day 2 at 760m and 3200m
  Difference in altitude-induced change (between day 2 at 760 meters a.s.l. vs. day 2 at 3200 meters a.s.l.) of center of gravity displacement between acetazolamide and placebo group, measured by a balance platform

SECONDARY OUTCOMES:
Change in arterial oxygen saturation | Day 2 at 760m and 3200m
  Difference in altitude-induced change (between day 2 at 760 meters a.s.l. vs. day 2 at 3200 meters a.s.l.) of arterial oxygen saturation between acetazolamide and placebo group, measured by pulse oximetry
acute mountain sickness | Day 2 at 3200m
  Difference in acute mountain sickness severity on day 2 at 3200 meters a.s.l. between acetazolamide and placebo group, measured by the environmental symptoms questionnaire cerebral subscore

CONTACTS AND LOCATIONS:
Overall Officials: Konrad E Bloch, MD, Study Chair — University of Zurich; Talant M Sooronbaev, MD, Study Director — National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan
Locations (1):
- National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan

IPD SHARING:
Plan to Share IPD: Undecided